CLINICAL TRIAL: NCT00985010
Title: Manganese, Possible Factor of Higher Mortality in Women With Encephalopathy
Brief Title: Manganese in Women With Encephalopathy
Status: Terminated | Type: Observational
Why Stopped: The authors finished their jobs in the hospitals where the study was begun.
Sponsor: Materno-Perinatal Hospital of the State of Mexico (Other)
Collaborators: Hospital General "Dr. Darío Fernández Fierro" (Unknown); National Institute of Neurology and Neurosurgery (Unknown)
Responsible Party: Hugo Mendieta Zerón, Materno-Perinatal Hospital of the State of Mexico
Other Study IDs: HGDrDFF-Mn2008
Record Dates: First submitted 2009-01-05; First posted 2009-09-25 (Estimated); Results first posted 2009-09-25 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2009-08

CONDITIONS: Hepatic Encephalopathy
Keywords: hepatic encephalopathy; hepatitis C; manganese; mortality; prognosis.
MeSH Terms: conditions — Hepatic Encephalopathy; Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective:

Report manganese serum levels and mortality in encephalopathic patients.

Patients and participants:

Consecutive patients aged > 18 years, with hepatic encephalopathy and informed consent signed by their families.

Interventions:

Patients' clinical characteristics as well as biochemical tests of renal function, hemoglobin, glucose and albumin levels were obtained as well as a blood sample to analyze manganese levels with a graphite furnace atomic absorption spectrometer.

Hypothesis:

There is a difference in the manganese levels between male and female patients.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients aged > 18 years
* With hepatic encephalopathy
* Informed consent signed by their families

Exclusion Criteria:

* Portal bypass surgery
* Cancer of any localization
* Known malignancy and other severe diseases which shorten life expectancy < 6 months
* Psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients aged > 18 years, with hepatic encephalopathy and informed consent signed by their families.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2003-01; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Mendieta Zerón, PhD, Principal Investigator — Materno-Perinatal Hospital of the State of Mexico; Camilo Rios Castañeda, PhD, Study Director — National Institute of Neurology and Neurosurgery; Mónica Rodríguez Rodríguez, MD, Study Chair — General Hospital "Dr. Darío Fernández Fierro"
Locations (1):
- General Hospital "Dr. Darío Fernández Fierro", México, D.f., Mexico

REFERENCES:
- [Derived] Zeron HM, Rodriguez MR, Montes S, Castaneda CR. Blood manganese levels in patients with hepatic encephalopathy. J Trace Elem Med Biol. 2011 Dec;25(4):225-9. doi: 10.1016/j.jtemb.2011.07.003. Epub 2011 Oct 4. PMID 21975221

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Encephalopathic patients admitted at the Department of Internal Medicine of the General Hospital "Dr. Darío Fernández Fierro" after being stabilized at the Emergency Room
Pre-assignment Details: They were consecutive patients males or females aged > 18 years, with hepatic encephalopathy.
Groups:
- Females; Males: Brain death
Period: Overall Study
Arm/Group | Females | Males
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Females | Males | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years]
  Between 18 and 65 years | 52.33 (3.05) | 56.66 (6.65) | 54.5 (5.2)
  >=65 years | 67 (0) | 72.5 (3.53) | 70.66 (4.04)
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (7.74) | 63 (10.02) | 59.88 (9.29)
Sex/Gender, Customized [Number; unit: participants]
  Between 18 and 65 years | 3 | 3 | 6
  >= 65 years | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  Mexico | 4 | 5 | 9
Baseline blood hemoglobin [Mean (Standard Deviation); unit: mg/dL] — Blood samples when arriving at the Emergency Room were used to measure hemoglobin
  mg/dL | 11.52 (1.57) | 12.14 (1.77) | 11.86 (1.61)
Blood levels of manganese [Mean (Standard Deviation); unit: µg/L] — Blood levels of manganese in patients with encephalopathy when arriving at the Emergency Room
  µg/L | 28.75 (9.47) | 18.5 (10.22) | 23.05 (10.72)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Evolution
Description: Number of participants who died versus those who remained alive after 6 months of follow up since the first entrance at the Emergency Room
Time Frame: six months
Population: We made a clinical follow up from nine encephalopathic patients. After six months we studied the differences in Mn, hemoglobin, etc., between those patients still alive and those who died.
Measure: Number; unit: participants
Arm/Group | Females | Males
Number analyzed (Participants) | 4 | 5
participants
  Still alive | 3 | 3
  deaths | 1 | 2
Statistical Analysis 1: Comparison: Females vs Males; Clinical evolution was reported as percentage (still alive or death after six months of follow up); Test type: Superiority or Other; p = 0.05, Chi-squared; Mean Difference (Final Values) = 15, Standard Deviation 5 — The difference is between the percentage of deaths (males versus females) after six months in the patients with hepatic encephalophathy

2. Secondary Outcome: Manganese Levels
Description: From encephalopathic patients, we took individual blood samples, analyzed in the biochemistry laboratory at the National Institute of Neurology and Neurosurgery, Mexico, City, with a graphite furnace atomic absorption spectrometer, according to the technique reported by Pleban.
Time Frame: Up to six months we followed the recruited patients to determine who were still alive
Population: All patients attended at the Internal Medicine Service with Hepatic Encephalopathy were included. The analysis was per protocol.
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Females | Males
Number analyzed (Participants) | 4 | 5
μg/L | 28.75 (9.4) | 18.5 (10.22)
Statistical Analysis 1: Comparison: Females vs Males; Laboratory results were expressed in means and standard deviations. Between group comparisons (female versus male values) were made with the Mann-Whitney U test using the Statistical Package for Social Sciences (SPSS) program version 10 (SPSS Inc., North Carolina, USA); Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 23.05, Standard Deviation 10.72 — The difference is between manganese levels of women minus manganese levels of men

ADVERSE EVENTS:
Arm/Group | Females | Males
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

LIMITATIONS AND CAVEATS:
Small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No